CLINICAL TRIAL: NCT05650008
Title: Effects of Intrathecal Local Anesthetics on Left Ventricular Global Longitudinal Strain
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Shayne Michael Roberts, Associate Professor, Department of Anesthesiology and Perioperative Medicine, Milton S. Hershey Medical Center
Other Study IDs: 21263
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Left Ventricular Dysfunction; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use; Global Cardiac Wall Motion Dysfunction
Keywords: Strain
MeSH Terms: conditions — Ventricular Dysfunction, Left; Sprains and Strains | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intrathecal local anesthesia — Administration of local anesthetic into intrathecal space to achieve surgical anesthesia
  Other Names: Spinal anesthesia

SUMMARY:
The objective of this study is to assess the effects of intrathecal local anesthetics on left ventricular global longitudinal strain (LVGLS) using transthoracic echocardiography (TTE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective knee and hip replacements under spinal anesthesia

Exclusion Criteria:

* Patients who do not wish to consent
* Patients with contraindications to TTE
* Patients with reduced left ventricular systolic function as defined by LV ejection fraction < 50% on pre-operative echocardiography
* Patients with body mass index greater than 40
* Non-English-speaking subjects
* Cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with no known history of LV dysfunction undergoing elective surgery under spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Global Longitudinal Strain | 5 minutes

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided